CLINICAL TRIAL: NCT02341846
Title: Exploring the Desirability, Feasibility and Practicalities of Using Information and Communication Technology (ICT) to Improve Cancer Pain Management in the Community
Brief Title: Exploring New Technologies to Manage Cancer Pain in the Community
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2/069/14
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-11

CONDITIONS: Neoplasms; Pain
Keywords: cancer pain
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with cancer pain: Qualitative semi-structured interviews with patients who have experienced cancer pain
  Interventions: Other: Qualitative interviews
- Caregivers for those with cancer pain: Qualitative semi-structured interviews with caregivers who have cared for those who have experienced cancer pain.
  Interventions: Other: Qualitative interviews
- Healthcare professionals: Healthcare professionals whose role involves the management of cancer pain.
  Interventions: Other: Qualitative interviews

INTERVENTIONS:
Other: Qualitative interviews

SUMMARY:
This interview and focus group study will explore patient, caregiver, and health professional opinions about the potential roles of digital technology to support effective cancer pain management. The views, opinions, and ideas expressed in this study will be used to design and develop a digital intervention which is likely to take the form of a measurement (pain and analgesic use) guided medication management intervention to improve cancer pain management in the community.

DETAILED DESCRIPTION:
Cancer is increasing in incidence and prevalence in the United Kingdom. Pain is the most frequent complication of cancer and cancer pain control is frequently suboptimal. Previous research has established several potentially modifiable reasons for suboptimal cancer pain management. These include: under-reporting of pain; inadequate communication about pain between patients and health care professionals ; inadequate assessment of pain by health care providers; inadequate analgesic prescribing; suboptimal adherence to prescribed analgesic regimens by patients; and failure to re-assess pain timeously.

Information and communication technology (ICT) is a term used to describe all digital technologies that facilitate the electronic capture, processing, storage, and exchange of information. ICT could offer innovative solutions to suboptimal cancer pain management. Technological solutions might include electronic diaries, available as applications or "apps", which could encourage pain self-monitoring by people with cancer, and prompt medical assessment when pain is poorly controlled. Accurate patient reported pain data could help professionals to adequately assess pain and might influence the patient-professional consultation. Feedback of adherence data to patients and carers might improve the way that medications are used. Electronic medication adherence devices are currently available which can capture data on analgesic utilisation and timing. This data might be useful for health care professionals to inform safe and timely adjustments of analgesic doses (i.e. is pain control poor because of inadequate analgesic dose or because of non-adherence to the prescribed regime?). The aim of the proposed study is to explore the desirability, feasibility, and practicalities of using ICT to improve cancer pain management The proposed study would seek the views of patients with cancer pain, their caregivers, and health care professionals, about using technology to help with cancer pain management. The study will investigate the acceptability of electronic pain diaries and electronic medication adherence devices to patients and health care professionals, barriers to using such technology, and how data generated from technology might be used by patients, caregivers, and health care professionals to improve cancer pain management. This study will form part of a programme of research and data from the proposed study will be used to inform the potential development of a technological intervention to improve the management of cancer pain in the community.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Adults, 18 years of age or over.
  * Established diagnosis of any cancer type.
  * Have experienced pain related to cancer or its treatment requiring any form of analgesic within the last three months.
  * Patients with all stages and grades of cancer who feel that they are willing and able to participate in an interview.

Caregivers • Caregivers aged 18 years of age or over who are or have been involved in providing care or assistance for somebody who has experienced cancer pain. Examples of caregivers might include family members, spouse, and close friends, who provide care and assistance to patients with cancer pain.

Professionals

• Registered doctors, nurses, and pharmacists who provide care for people with cancer pain.

Exclusion Criteria:

* • Non- English language speakers. Qualitative investigations will be reliant on communication in English. Specific words and phrases will be analysed by English speaking researchers in order to identify thematic content. This study does not include resources for interpreting services.

  * Patients who are thought to have entered the terminal stages of their illness will be excluded. This will be judged at recruitment by the screening clinician from the patient's general practice. In the case that a recruited patient has become too ill to participate in the research or has died before participation, and a linked caregiver has expressed interest in the study, the caregiver will be contacted, offered sympathies, and will be given the opportunity to withdraw from the study or continue as planned. All conversations about the study will be conducted in a supportive manner that recognises the sensitivity of the subject matter.
  * Patients who are registered at Great Western Medical Practice, Aberdeen (Rosalind Adam, researcher and interviewer practices as a doctor there).
  * Any participant who declines to take part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer pain, their caregivers, and health care professionals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Qualitative semi-structured interviews | Eight months

REFERENCES:
- [Derived] Adam R, Bond CM, Burton CD, de Bruin M, Murchie P. Can-Pain-a digital intervention to optimise cancer pain control in the community: development and feasibility testing. Support Care Cancer. 2021 Feb;29(2):759-769. doi: 10.1007/s00520-020-05510-0. Epub 2020 May 28. PMID 32468132